CLINICAL TRIAL: NCT05230069
Title: Assessment of a Prehospital Mobile App and Sensor Triage System to Detect Neurologic and Cardiac Emergencies: The ECHAS Assessment Study (ECHAS- One)
Brief Title: Emergency Call for Heart Attack and Stroke (ECHAS) - ECHAS One Study
Acronym: ECHAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Emergency Call for Heart Attack and Stroke (ECHAS) (Industry)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Sponsor
Other Study IDs: ECHAS One
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Heart Attack and Stroke
Keywords: Triage; Smartphone
MeSH Terms: conditions — Myocardial Infarction; Stroke | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients post emergency evaluation: Interview of patients post notification of emergency system
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed post an emergency call and evaluation.

SUMMARY:
ECHAS One will test the use of a smartphone app to assist patients to decide if it is necessary to call for emergency care with symptoms that could represent a heart attack or stroke.

DETAILED DESCRIPTION:
The ECHAS One Study will be conducted in 200 patients who have already called for emergency care for a heart or stroke, and have been evaluated. The endpoint of the study will be a decision if the initial call was an appropriate call for emergency care. The sensitivity of the app for detecting appropriate calls will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Presented to ED via emergency medical services (EMS) for "Stroke alert" symptoms, including:

Slurred speech Asymmetric weakness or numbness Balance problems Vision changes Headache

And/or "MI alert" symptoms including:

Chest discomfort Chest pressure or pain Palpitations Shortness of breath Lightheadedness or presyncope Syncope Age ≥ 18 years Able to provide informed consent

Exclusion Criteria:

* Non-English speaking
* Moderate or greater dementia
* Severe visual impairment
* Inability to use smartphone (for physical, cognitive, or other reasons)
* Unable to consent for study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 200 patients who activated emergency system for symptoms of possible heart attack or stroke.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Appropriate Emergency Activation | 3 months
  Was the right call made for a possible heart attack or stroke

CONTACTS AND LOCATIONS:
Overall Officials: James E Muller, Study Director — CEO, ECHAS, LLC

IPD SHARING:
Plan to Share IPD: No